CLINICAL TRIAL: NCT03386032
Title: 8-Week Atopic Dermatitis (AD) Treatment Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSD2017168
Record Dates: First submitted 2017-12-15; First posted 2017-12-29 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Atopic Dermatitis Eczema
MeSH Terms: interventions — Desonide

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized and balanced into one of the 3 treatment groups by their baseline SCORAD grade (moderate = 25-40 and severe = 41+) and ethnicity (black or non-black).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: As above
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Investigational OTC Cream (Experimental): Investigational Over the Counter (OTC) Cream will be applied topically, twice daily, for 8 weeks, once in the morning and once in the evening, to atopic dermatitis lesions and whole body as moisturizer.
  Interventions: Drug: Investigational OTC Cream
- Placebo Cream (Sham Comparator): Placebo Cream will be applied topically, twice daily, for 8 weeks, once in the morning and once in the evening, to atopic dermatitis lesions and whole body as body moisturizer.
  Interventions: Other: Placebo Cream
- 0.05% Desonide Cream (Active Comparator): Rx Steroid applied topically, twice daily, once in the morning and once in the evening, for 8 weeks to all atopic dermatitis lesions.
  Placebo Cream applied topically, twice daily, for 8 weeks, once in the morning and once in the evening, to whole body as body moisturizer, except atopic dermatitis lesions.
  Interventions: Drug: 0.05% Desonide; Other: Placebo Cream

INTERVENTIONS:
Drug: Investigational OTC Cream — Investigational Over the Counter (OTC) Cream applied topically, twice daily, for 8 weeks, once in the morning and once in the evening, to atopic dermatitis lesions and whole body as moisturizer.
  Arms: Investigational OTC Cream
Drug: 0.05% Desonide — Rx Steroid applied topically, twice daily, once in the morning and once in the evening, for 8 weeks to all atopic dermatitis lesions.
  Placebo Cream applied topically, twice daily, for 8 weeks, once in the morning and once in the evening, to whole body as body moisturizer, except atopic dermatitis lesions.
  Other Names: Desowen
  Arms: 0.05% Desonide Cream
Other: Placebo Cream — Placebo Cream applied topically, twice daily, for 8 weeks, once in the morning and once in the evening, to atopic dermatitis lesions and whole body as body moisturizer.
  Other Names: Vehicle
  Arms: 0.05% Desonide Cream; Placebo Cream

SUMMARY:
This is a study to investigate the clinical effectiveness of the Sponsor's experimental cream treatment on eczema as measured by visual grading of SCORAD (scoring of atopic dermatitis).

DETAILED DESCRIPTION:
This will be a 9-week, randomized, double blind, parallel comparison study consisting of a 1-week washout phase followed by an 8-week treatment phase. This study will be executed by one clinical research company utilizing two test sites and up to 62 subjects with moderate or severe atopic dermatitis, ages 12-65, will be enrolled. Subjects that are enrolled will be placed on one of three products (e.g. Sponsor's Experimental Cream Treatment, a basic moisturizer, or a positive control - Desonide) and will be required to use the assigned product twice a day for the duration of the 8-week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Is a generally healthy, male or female, 12-65 years old, inclusive;
* Diagnosis of moderate or greater Atopic Dermatitis as determined by SCORAD (SCORAD >=25);
* Is able to read and understand instructions in English.

Exclusion Criteria:

* Is currently participating or has participated in another interventional clinical study in the past 2 weeks;
* Currently or has been diagnosed or treated for cancer in the past 5 years;
* Requires any topical or systemic medications that could affect the course of their atopic dermatitis during the study period (except inhaled steroids and/or stable antihistamines for asthma or allergies);
* Has used systemic treatments that could affect AD within 30 days or 5 half- lives. (i.e. retinoids, methotrexate, cyclosporine, hydroxycarbamide (hydroxyurea), azathioprine and oral/injectable corticosteroids);
* Has a known hypersensitivity to any corticosteroid creams;
* Has been diagnosed with any allergies to Oat or derivatives;
* Has any active infections or has used antibiotics in the past 7 days;
* Has any physical attributes or skin conditions that might interfere with the clear visual or instrumental assessments.(i.e. cuts, sunburn, birth marks, tattoos, extensive scarring, excessive hair growth or acne);
* Has an immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus rheumatoid arthritis) which could place the subject at risk or interfere with the accuracy of the study results;
* Has used any immunosuppressant drugs or immunotherapy within the past 30days or 5 half-lives;
* Is an employee of the sponsor company or clinical testing site;
* Is diabetic;
* Presents with the presence of an active or chronic allergic reaction as evidenced by an irregular white cell count determined by eosinophils > 0.3 X 109/L at Screening Visit;
* Is planning a trip to a sunny climate, to use tanning booths or use other UV sources throughout the course of this study;
* Has a history of hypersensitivity to any substance in investigational preparation or to Desonide;
* Has any clinically significant medical condition or laboratory abnormality that would, in the opinion of the Investigator, put the patient at undue risk or interfere with the interpretation of the study results;
* Is dependent on oral medication for any skin disease/condition or could not, in the opinion of the Investigator tolerate the restriction of discontinuing the medicine as required in this study;
* Is currently pregnant or lactating or planning to become pregnant in the next 6 months;
* Has other skin conditions that might interfere with AD diagnosis and/or evaluation (i.e. psoriasis current active viral, bacterial and fungal skin infections) as assessed by the Investigator;
* Any other condition or factor the Investigator or their duly assigned representative believes may affect the ability of the subject to complete the study or the interpretation

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Salisbury, BSN, Study Director — Wake Research, LLC
Locations (2):
- United States (2):
  - Wake Research, LLC, Raleigh, North Carolina
  - WR (Wake Research) ClinSearch, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.05% Desonide Cream: Rx Steroid applied topically, twice daily, once in the morning and once in the evening, for 8 weeks to all atopic dermatitis lesions.
  Placebo Cream applied topically, twice daily, for 8 weeks, once in the morning and once in the evening, to whole body as body moisturizer, except atopic dermatitis lesions.
  0.05% Desonide: Rx Steroid applied topically, twice daily, once in the morning and once in the evening, for 8 weeks to all atopic dermatitis lesions.
  Placebo Cream applied topically, twice daily, for 8 weeks, once in the morning and once in the evening, to whole body as body moisturizer, except atopic dermatitis lesions.
  Placebo Cream: Placebo Cream applied topically, twice daily, for 8 weeks, once in the morning and once in the evening, to atopic dermatitis lesions and whole body as body moisturizer.
Period: Overall Study
Arm/Group | Investigational OTC Cream | Placebo Cream | 0.05% Desonide Cream
Started | 36 | 18 | 11
Completed | 18 | 11 | 11
Not Completed | 18 | 7 | 0
Not completed — Lack of Efficacy | 6 | 2 | 0
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 9 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational OTC Cream | Placebo Cream | 0.05% Desonide Cream | Total
Number analyzed (Participants) | 36 | 18 | 11 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (13.5) | 39.6 (15.3) | 42 (15.4) | 37.3 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 15 | 7 | 47
  Male | 11 | 3 | 4 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 9 | 6 | 31
  White | 19 | 9 | 4 | 32
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 18 | 11 | 65
SCORAD [Mean (Standard Deviation); unit: units on a scale] — SCORAD (Severity Scoring of Atopic Dermatitis) is a composite severity index comprising:
  * Extent (a) of body area affected [graded 0-100];
  * Objective (b) assessments on the intensity of symptoms of Dryness/Scaling, Erythema, Excoriation, Induration/Papulation, Lichenification and Oozing/Weeping/Crusting, [each graded from 0 (None) to 3 (Severe)]
  * Subjective (c) assessment of Itch and Sleep Disturbance, graded via 10 pt visual analog assessments
  SCORAD is calculated as a/5 + 3.5*b + c, with totals ranging from 0 (No Atopic Dermatitis) to 103 (Severe). A Lower SCORAD # is Better.
  units on a scale | 49.18 (2.39) | 52.21 (3.36) | 45.22 (4.33) | 49.3 (14.1)

OUTCOME MEASURES:

1. Primary Outcome: Severity Scoring of Atopic Dermatitis (SCORAD) Amongst Subjects With Moderate Atopic Dermatitis
Description: SCORAD (Severity Scoring of Atopic Dermatitis) Change from Baseline to Week 8 of atopic dermatitis lesion as measured by the Scoring of Atopic Dermatitis (SCORAD). SCORAD is a composite severity index comprising a) the amount/extent of body area affected; b)b) 2 subjective symptom of pruritus (10 pts VAS) and sleep disturbance measured (10 pts VAS); and c) 6 disease intensity assessments [Dryness/Scaling, Erythema, Excoriation, Induration/Papulation, Lichenification and Oozing/ Weeping/Crusting, each graded in 3pts TIS from 0 (None) to 3 (Severe). A SCORAD score ranges from 0 (No AD present) to 103
  SCORAD is calculated:
  Extent 7*Intensity SCORAD = --------- + ---------------- + Subjective 5 2
Time Frame: Baseline to Week 8
Population: Subjects with moderate Atopic Dermatitis as defined by Baseline SCORAD 25-40
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Investigational OTC Cream | Placebo Cream | 0.05% Desonide Cream
Number analyzed (Participants) | 11 | 4 | 3
units on a scale | -12.2 (3.99) | 9.3 (6.51) | -17.5 (8.29)
Statistical Analysis 1: Comparison: Investigational OTC Cream vs Placebo Cream vs 0.05% Desonide Cream; Change from baseline in variables were analyzed separately using a mixed model for repeated measures with Subject nested within treatment (random effect), and Treatment, Week, Treatment-by-Week, Age & Baseline (fixed effects). Last Observation was Carried Forward (LOCF) for drops. Sporadic missing data were left missing; Test type: Superiority; p < 0.05, ANCOVA; Model adjusted means

2. Primary Outcome: Severity Scoring of Atopic Dermatitis (SCORAD) Amongst Subjects With Severe Atopic Dermatitis
Description: as for outcome 1
Time Frame: Baseline to Week 8
Population: Subjects with severe Atopic Dermatitis (Baseline SCORAD = 41+)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Investigational OTC Cream | Placebo Cream | 0.05% Desonide Cream
Number analyzed (Participants) | 19 | 11 | 7
units on a scale | -6.0 (2.8) | -20.3 (3.7) | -18.0 (4.5)
Statistical Analysis 1: Comparison: Investigational OTC Cream vs Placebo Cream vs 0.05% Desonide Cream; Change from baseline in variables were analyzed separately using a mixed model for repeated measures with Subject nested within treatment (random effect), and Treatment, Week, Treatment-by-Week, Age & Baseline (fixed effects). Last Observation was Carried Forward (LOCF) for drops. Sporadic missing data were left missing. Significance level: 0.05 (2-sided); Test type: Superiority; p < 0.05, ANCOVA; Model adjusted means. Last Observation was Carried Forward (LOCF) for drops. Sporadic missing data were left miss

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the subject's participation in the study (up to 8 weeks).
Arm/Group | Investigational OTC Cream | Placebo Cream | 0.05% Desonide Cream
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/18 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/18 | 0/11
Other Adverse Events (participants affected / at risk) | 2/36 | 2/18 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational OTC Cream (N=36) | Placebo Cream (N=18) | 0.05% Desonide Cream (N=11)
Atopic /Other (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is employed by a contract research organization that is solely responsible for execution of the protocol. The contract research organization (and the PI) have signed a non-disclosure agreement, agreeing to keep all study-related information confidential. The Sponsor is responsible for data analysis.

DOCUMENTS (2):
  • Study Protocol (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03386032/Prot_002.pdf
  • Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03386032/SAP_003.pdf